CLINICAL TRIAL: NCT00543088
Title: SERENITY: Evaluating the Effectiveness of Atypical Antipsychotics in the Community - a Prospective, Multicentre, Observational Study to Evaluate the Impact on Quality of Life of GP-Bases Management of Antipsychotic Treatment in Belgium.
Brief Title: Effectiveness of Anti-Psychotic in GPs Setting
Acronym: Serenity
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: SRP-NB-SER-2006/1
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; Bipolar Disorder; manic episode; atypical antipsychotic; Schizophrenia or Bipolar Disorder (currently in a manic episode)
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Mania

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluating the effectiveness of atypical antipsychotics in the community - a prospective, multicentre, observational study to evaluate the impact on Quality of Life of GP-based management of antipsychotic treatment in Belgium

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Schizophrenia or Bipolar Disorder (currently in a manic episode)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2007-01; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
to evaluate the patient's functioning, by measuring the Quality of Life. Quality of Life will be assessed by the Q-LES-Q-16 (PRO).

SECONDARY OUTCOMES:
The clinical efficacy & tolerability of atypical antipsychotics as assessed by the Clinical Global Impression(CGI) & Patient Global Impression of Change(PGIC)scores.
The wellbeing of the patients taking atypical antipsychotics as assessed by the Sheehan Disability Scale(SDS)

CONTACTS AND LOCATIONS:
Overall Officials: Pitchot W Pr, Principal Investigator — ULg
Locations (57):
- Belgium (57):
  - Research Site, Baudour
  - Research Site, Beyne-Heysay
  - Research Site, Bomal
  - Research Site, Bredene
  - Research Site, Brussels
  - Research Site, Esen
  - Research Site, Evere
  - Research Site, Gingelom
  - Research Site, Gouy-lez-Piéton
  - Research Site, Grâce-Hollogne
  - Research Site, Gullegem
  - Research Site, Harelbeke
  - Research Site, Harre
  - Research Site, Hotton
  - Research Site, Houtvenne
  - Research Site, Incourt
  - Research Site, Ixelles-Elsene
  - Research Site, Jalhay
  - Research Site, Jette
  - Research Site, Keumiée
  - Research Site, Lembeke
  - Research Site, Liège
  - Research Site, Limbourg
  - Research Site, Longueville
  - Research Site, Lovendegem
  - Research Site, Malmedy
  - Research Site, Mechelen
  - Research Site, Monceau-sur-Sambre
  - Research Site, Montignies-sur-Sambre
  - Research Site, Moorsel
  - Research Site, Moorseled
  - Research Site, Mouscron
  - Research Site, Namur
  - Research Site, Oostrozebeke
  - Research Site, Ostend
  - Research Site, Oudenaarde
  - Research Site, Poperinge
  - Research Site, Ransart
  - Research Site, Roux
  - Research Site, Ruisbroek
  - Research Site, Schaarbeek
  - Research Site, Spa
  - Research Site, Staden
  - Research Site, Theux
  - Research Site, Tilleur
  - Research Site, Torhout
  - Research Site, Tubize
  - Research Site, Verviers
  - Research Site, Veurne
  - Research Site, Wachtebeke
  - Research Site, Willebroek
  - Research Site, Wilrijk
  - Research Site, Woluwe-St-Lambert
  - Research Site, Zeebrugge
  - Research Site, Zichem
  - Research Site, Zomergem
  - Research Site, Zonnebeke